CLINICAL TRIAL: NCT03102710
Title: Neuromodulation of Placebo and Nocebo Effects
Brief Title: Neuromodulation of Lidocaine and Capsaicin Cream Effects on Pain Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015P000685
Record Dates: First submitted 2017-01-27; First posted 2017-04-06 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- tDCS Enhancement (Experimental): In this group, the transcranial direct current stimulation (tDCS) stimulates the areas of the brain being examined in this study to increase their activity.
  Interventions: Device: transcranial direct current stimulation (tDCS); Other: Lidocaine cream; Other: Capsaicin cream; Other: Control cream
- tDCS Inhibition (Experimental): In this group, the transcranial direct current stimulation (tDCS) inhibits the areas of the brain being examined in this study to decrease their activity.
  Interventions: Device: transcranial direct current stimulation (tDCS); Other: Lidocaine cream; Other: Capsaicin cream; Other: Control cream
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation (tDCS) does not provide real stimulation though you will not know this until your debriefing at the end of the study. Sham will be used to determine if the results of this study are due to the tDCS or other reasons.
  Interventions: Device: transcranial direct current stimulation (tDCS); Other: Lidocaine cream; Other: Capsaicin cream; Other: Control cream

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tCDS safely applies a weak electrical current to your scalp using two sponge electrodes that look like flat circular pads. The pads will be held in place on your head with a neoprene cap. The pads will be attached to a generator that will send a weak stimulus to your scalp. This current influences the way that your brain cells work. When the stimulus starts, you might feel a tingling sensation underneath the electrode pads. That sensation is not painful and goes away in seconds.
Other: Lidocaine cream — Lidocaine cream will be applied on the arm to reduce pain sensitivity (analgesia).
Other: Capsaicin cream — Capsaicin cream will be applied on the arm to increase pain sensitivity (hyperalgesia).
Other: Control cream — A neutral cream will be applied on the arm as a control.

SUMMARY:
The aim of this study is to use a brain stimulation tool called transcranial direct current stimulation (tDCS) to investigate the analgesic (reducing sensitivity to pain) effects of lidocaine cream and the hyperalgesic (increasing sensitivity to pain) effects of capsaicin cream using a neutral cream as a control. tDCS stimulation has been shown to temporarily influence the way the stimulated part of the brain functions. With this method, the involvement of specific parts of the brain can be investigated in the working of the brain as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Right handed healthy male and female adults aged 21-50
* No contraindications to fMRI scanning
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Current or past history of major medical, neurological, or psychiatric illness
* Claustrophobia
* History of head trauma
* Instability of responses to experimental pain
* Non-fluent speaker of English
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy
* History of alcohol/substance abuse

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 subjects were dropped prior to randomization. Reasons for this included inconsistent or non-differentiable pain ratings to heat stimuli, pain thresholds that were too high or low, inability to finish subsequent sessions, too much discomfort with noxious stimuli, no SSN/hairstyle incompatible with tDCS, participated in a previous pain study.
Groups:
- Sham tDCS: Sham transcranial direct current stimulation (tDCS) does not provide real stimulation though you will not know this until your debriefing at the end of the study. Sham will be used to determine if results of this study are due to tDCS or other reasons.
  transcranial direct current stimulation (tDCS): tCDS safely applies a weak electrical current to your scalp using two sponge electrodes that look like flat circular pads. The pads will be held in place on your head with a neoprene cap. The pads will be attached to a generator that will send a weak stimulus to your scalp. This current influences the way that your brain cells work. When the stimulus starts, you might feel a tingling sensation underneath the electrode pads. That sensation is not painful and goes away in seconds.
  Lidocaine cream: Lidocaine cream will be applied on the arm to reduce pain sensitivity (analgesia).
  Capsaicin cream: Capsaicin cream will be applied on the arm to increase pain sensitivity (hyperalgesia).
Period: Overall Study
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS
Started | 28 | 30 | 27
Completed | 27 | 27 | 27
Not Completed | 1 | 3 | 0
Not completed — Dental metal affected MRI scan quality | 1 | 0 | 0
Not completed — Technical issues during final MRI scan | 0 | 1 | 0
Not completed — Nausea during MRI scan | 0 | 1 | 0
Not completed — Subject unable to attend final session | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed all study sessions
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS | Total
Number analyzed (Participants) | 27 | 27 | 27 | 81
Age, Continuous [Mean (Full Range); unit: years] | 27.42 [21.40 to 47.39] | 26.87 [21.09 to 47.19] | 27.89 [21.25 to 49.23] | 27.39 [21.09 to 49.23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 13 | 37
  Male | 14 | 16 | 14 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 3 | 13
  Not Hispanic or Latino | 20 | 21 | 23 | 64
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 4 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 6
  White | 18 | 19 | 15 | 52
  More than one race | 2 | 0 | 5 | 7
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 27 | 81
Baseline pain ratings for low pain stimuli [Mean (Standard Deviation); unit: units on a scale] — The Gracely Sensory Scale, which ranges from 0-20, is used to rate pain experiences. 0 indicates no pain sensation, and 20 indicates extremely intense pain.
  units on a scale | 6.05 (2.67) | 4.54 (2.04) | 5.08 (2.14) | 5.22 (2.36)
Baseline pain ratings for moderate pain stimuli [Mean (Standard Deviation); unit: units on a scale] — The Gracely Sensory Scale, which ranges from 0-20, is used to rate pain experiences. 0 indicates no pain sensation, and 20 indicates extremely intense pain.
  units on a scale | 9.31 (1.97) | 8.84 (2.54) | 8.97 (2.34) | 9.04 (2.28)
Baseline pain ratings for high pain stimuli [Mean (Standard Deviation); unit: units on a scale] — The Gracely Sensory Scale, which ranges from 0-20, is used to rate pain experiences. 0 indicates no pain sensation, and 20 indicates extremely intense pain.
  units on a scale | 14.52 (2.67) | 14.56 (2.33) | 14.52 (2.20) | 14.53 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Functional Connectivity Changes of the DLPFC Before and After tDCS Stimulation
Description: We investigated the effects of cathodal (inhibition) and anodal (enhancement) tDCS on rDLPFC functional connectivity (FC) with the supplementary motor area (SMA) and anterior insula. Higher Fisher Z-scores represent greater resting-state functional connectivity.
Time Frame: up to 2 weeks
Population: Participants who completed all study sessions
Measure: Mean (Standard Deviation); unit: Fisher Z value
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS
Number analyzed (Participants) | 27 | 27 | 27
Fisher Z value
  rDLPFC-SMA Functional Connectivity (post-pre) | -0.11 (0.22) | -0.09 (0.16) | 0.08 (0.20)
  rDLPFC-Insula Functional Connectivity (post-pre) | -0.13 (0.23) | -0.13 (0.20) | 0.07 (0.18)

2. Primary Outcome: fMRI Resting States Functional Connectivity Changes During Pain Stimulation
Description: We measured changes in blood oxygen level-dependent (BOLD) activity in the brain during pain stimulation. In the outcome measure data table, "placebo contrast" indicates lidocaine - neutral and "nocebo contrast" indicates capsaicin - neutral.
Time Frame: up to 2 weeks
Population: Participants who completed all study sessions and whose task fMRI data had no issues.
Measure: Mean (Standard Deviation); unit: Arbitrary unit
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS
Number analyzed (Participants) | 26 | 27 | 26
Arbitrary unit
  BOLD activity change in mPFC/ACC: placebo contrast | 0.14 (0.47) | 0.50 (0.57) | -0.17 (0.68)
  BOLD activity change in mPFC/ACC: nocebo contrast | 0.26 (0.80) | 0.27 (0.81) | 0.25 (1.15)
  BOLD activity in the left insula: placebo contrast | 0.11 (0.35) | 0.21 (0.81) | 0.18 (0.64)
  BOLD activity in the left insula: nocebo contrast | 0.08 (0.36) | 0.16 (0.35) | 0.30 (0.39)

3. Secondary Outcome: Gracely Sensory Scale Pain Rating Changes in Response to Lidocaine and Capsaicin Creams and tDCS
Description: The Gracely Sensory Scale allows participants to rate the intensity of heat pain stimuli on a scale from 0 to 20, with 0 indicating no pain sensation and 20 indicating extremely intense pain. The outcome measure data table shows mean pain ratings for the lidocaine, capsaicin, and neutral creams after enhancement, inhibition, or sham tDCS stimulation.
Time Frame: up to 2 weeks
Population: Participants who completed all study sessions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS
Number analyzed (Participants) | 27 | 27 | 27
units on a scale
  Pain rating on nocebo cream | 8.54 (3.54) | 8.80 (2.60) | 9.01 (2.75)
  Pain rating on placebo cream | 7.29 (2.74) | 6.41 (2.86) | 7.38 (2.84)
  Pain rating on neutral cream | 8.10 (2.65) | 7.96 (2.90) | 7.88 (2.56)
Statistical Analysis 1: Comparison: tDCS Enhancement vs tDCS Inhibition vs Sham tDCS; To assess the modulation effects of tDCS on placebo, we first performed an analysis of covariance (ANCOVA) with placebo as the dependent variable and group (i.e., anodal, cathodal, and sham tDCS) as the fixed factor; Test type: Superiority — Covariates included 1) age, 2) cream randomization, and 3) the difference in ERS for lidocaine before and after expectancy manipulation (which represented how well the expectancy was modulated) in Session 2; p = 0.03, ANCOVA — The threshold for significance was <0.05; Mean Difference (Final Values) = 0.4 — The mean difference between anodal vs. sham was 0.4, between cathodal vs. sham was 1.2, and between anodal vs. cathodal was -0.8
Statistical Analysis 2: Comparison: tDCS Enhancement vs tDCS Inhibition vs Sham tDCS; To assess the modulation effects of tDCS on nocebo, we first performed an analysis of covariance (ANCOVA) with nocebo as the dependent variable and group (i.e., anodal, cathodal, and sham tDCS) as the fixed factor; Test type: Superiority — Covariates included 1) age, 2) cream randomization, and 3) the difference in ERS for capsaicin before and after expectancy manipulation (which represented how well the expectancy was modulated) in Session 2. In addition, we added the STAI state and trait anxiety scores as covariates when assessing the modulation effects of tDCS on the nocebo effect, as previous studies have suggested that anxiety level could affect nocebo hyperalgesia; p = 0.04, ANCOVA — The threshold for significance was <0.05; Mean Difference (Final Values) = 1.3 — The mean difference between anodal vs. sham was 1.4, between cathodal vs. sham was 1.0, and between anodal vs. cathodal was -0.3

ADVERSE EVENTS:
Time Frame: Up to 2 weeks for each participant (during participation in the study)
Description: The occurrence of adverse events were assessed by study staff at each site visit. Adverse events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | tDCS Enhancement | tDCS Inhibition | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 2/28 | 1/30 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS Enhancement (N=28) | tDCS Inhibition (N=30) | Sham tDCS (N=27)
Unpleasant tDCS Sensations (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Complaints of unpleasant tDCS sensations during MRI scan.
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Participant complained of nausea during MRI scan

LIMITATIONS AND CAVEATS:
The sample size for this study was relatively small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT03102710/ICF_000.pdf
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03102710/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03102710/SAP_002.pdf